CLINICAL TRIAL: NCT05702372
Title: Short-term Effects of Crackers on Glycemic Index and Glycemic Responses. A Randomized Trial in Healthy Adults
Brief Title: Acute Glycemic Effects of Crackers Made by Different Flours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Collaborators: Institute of Technology and Agricultural Products (Unknown)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HRBD 80/12.10.2022
Record Dates: First submitted 2023-01-19; First posted 2023-01-27 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetitive Behavior
Keywords: blood glucose; crackers; glycemic index; glycemic load
MeSH Terms: conditions — Appetitive Behavior | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Crossover assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: double-blind (investigator and outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Glucose as reference food (Experimental): Eleven healthy, normal body weight adults (male: 4, female: 7) after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g of available carbohydrates from crackers made by wheat, rye and sunflower flours, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food
- Cracker made by wheat flour (Experimental): Eleven healthy, normal body weight adults (male: 4, female: 7) after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g of available carbohydrates from crackers made by wheat, rye and sunflower flours, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Cracker made by wheat flour
- Cracker made by rye flour (Experimental): Eleven healthy, normal body weight adults (male: 4, female: 7) after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g of available carbohydrates from crackers made by wheat, rye and sunflower flours, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Cracker made by rye flour
- Cracker made by sunflower flour (Experimental): Eleven healthy, normal body weight adults (male: 4, female: 7) after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g of available carbohydrates from crackers made by wheat, rye and sunflower flours, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Cracker made by sunflower flour

INTERVENTIONS:
Other: Glucose as reference food — Eleven healthy, normal weight subjects after 10-14 hours fast, consumed 50g glucose diluted in 300ml water, tested three times, in different visits, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
  Arms: Glucose as reference food
Other: Cracker made by wheat flour — Eleven healthy, normal weight subjects after 10-14 hours fast, consumed 50g available carbohydrates from cracker made by wheat flour, along with 300ml water, tested once, within 10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
  Arms: Cracker made by wheat flour
Other: Cracker made by rye flour — Eleven healthy, normal weight subjects after 10-14 hours fast, consumed 50g available carbohydrates from cracker made by rye flour, along with 300ml water, tested once, within 10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
  Arms: Cracker made by rye flour
Other: Cracker made by sunflower flour — Eleven healthy, normal weight subjects after 10-14 hours fast, consumed 50g available carbohydrates from sunflower flour, along with 300ml water, tested once, within 10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
  Arms: Cracker made by sunflower flour

SUMMARY:
This study investigated the acute effects of cracker consumption made by different flours on glycemic responses.

DETAILED DESCRIPTION:
This study aimed to determine the glycemic index and glycemic load of crackers made by different flours (wheat, whole wheat, and 30% sunflower seed flour substitution) and to investigate the effects of these types of crackers on postprandial glycemic responses in healthy humans. Moreover, blood pressure levels and subjective appetite were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking
* non-diabetic men and women
* body mass index between 18 and 25 kg/m2

Exclusion Criteria:

* severe chronic diseases (e.g. cardiovascular diseases, diabetes mellitus, kidney or liver conditions, endocrine conditions)
* gastrointestinal disorders
* pregnancy
* lactation
* competitive sports
* alcohol abuse
* drug dependency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Glycemic index | 2 hours
  Glucose solution (50 g) was the reference food (GI = 100%) against which all test foods were compared. Subjects arrived at the laboratory at eight to nine o'clock in the morning after 10-12 h overnight fast. Each subject was fed equivalent 50 g available carbohydrate of test foods or reference food in random order. To minimize day to day variation of glucose tolerance, the reference food was tested in triplicate in each subject. All test and reference foods were served with 250 mL of water. An automatic lancet device and glucometer (calibrated MediSmart Ruby glucose meter with a lancing device, Lilly-PHARMASERV SA, Greece) was used for finger capillary blood samples. Blood samples were taken immediately before the start of the study (0 min) and 15, 30, 45, 60, 90 and 120 min after the start of eating.
Capillary blood glucose responses | 2 hours
  Clinically useful change in blood glucose, defined as the restoration of glucose within normal limits during the 2hr glucose tolerance test

SECONDARY OUTCOMES:
Subjective appetite ratings | 2 hours
  Useful change in subjective appetite using visual analogue scales with a score 0 to 10 (given in the form of booklet, one scale per page) at baseline, 15, 30, 45, 60, 90 and 120min. The minimum or maximum score will be evaluated if it is better or worse depending on the appetite variable e.g. hunger, satiety, desire to eat etc
Blood pressure | 2 hours
  Useful change in systolic and diastolic blood pressure before and 2hr after consumption of the spaghetti productws

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papakonstantinou E, Alsab V, Lympaki F, Chanioti S, Giannoglou M, Katsaros G. The acute effects of variations in the flour composition of crackers on the glycemic index and glycemic responses in healthy adults. Eur J Clin Nutr. 2024 Dec;78(12):1051-1057. doi: 10.1038/s41430-024-01482-0. Epub 2024 Aug 5. PMID 39103546